CLINICAL TRIAL: NCT05337566
Title: Infections After Hysterectomy - a Placebo-controlled Study Comparing the Prophylactic Use of Azithromycin and Cefuroxime With Single Cefuroxime
Brief Title: Does Additional Use of Preoperative Azithromycin Decrease Posthysterectomy Infections
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: University of Turku (Other); Tampere University Hospital (Other); Kuopio University Hospital (Other); Oulu University Hospital (Other); Jyväskylä Central Hospital (Other)
Responsible Party: Principal Investigator, Päivi Rahkola-Soisalo, Adjuct professor, M.D., Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HUS/117/2022; 2021-003467-10 (EudraCT Number)
Record Dates: First submitted 2022-04-14; First posted 2022-04-20 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Infection Post Op; Hysterectomy; Antibiotics; Prophylactic
Keywords: postoperative, infection, hysterectomy, antibiotics
MeSH Terms: conditions — Infections | interventions — Azithromycin; Cefuroxime

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: single blinded - the placebo tablets slightly differ from the azithromycin tablets, therefore they are sealed in package which is given straight to the participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Azithromycin + Cefuroxime (Experimental): Changed with renewed study permissions:
  These patients will receive Azithromycin 500 mg (2 tablets) per orally on the operation day when they arrive to the hospital and a single dose Cefuroxime 1.5g (when body mass index is under 30) or 3g (for those whose bosy mass index is 30 or more) in the operating theatre before the incision.
  The previous description:
  These patients will receive Azithromycin 500 mg (2 tablets) per orally in the evening before the operation and single dose Cefuroxime 1.5g (when body mass index is under 30) or 3g (for those whose body mass index is 30 or more) in the operating theatre before the incision.
  Interventions: Drug: Azithromycin Pill + Cefuroxime
- Placebo + Cefuroxime (Active Comparator): Changed with new study permissions:
  These patients will receive placebo (2 tablets) per orally on the operation day when they arrive to the hospital and a single dose Cefuroxime 1.5g (when body mass index is under 30) or 3g (for those whose bosy mass index is 30 or more)in the operating theatre before the incision.
  The previous description:
  These patients will receive placebo (2 tablets) per orally in the evening before the operation and a single dose Cefuroxime 1.5g (when body mass index is under 30) or 3g (for those whose body mass index is 30 or more) in the operating theatre before the incision.
  Interventions: Drug: Placebo + Cefuroxime

INTERVENTIONS:
Drug: Azithromycin Pill + Cefuroxime — Azithromycin 500 mg (2 tablets) per orally when arriving to the hospital before the operation and a single dose Cefuroxime 1.5g (when body mass index is under 30) or 3g (for those whose body mass index is 30 or more) in the operating theatre before the incision
  Arms: Azithromycin + Cefuroxime
Drug: Placebo + Cefuroxime — Placebo (2 tablets) per orally in the evening when arriving to the hospital before the operation and a single dose Cefuroxime 1.5g (when body mass index is under 30) or 3g (for those whose body mass index is 30 or more) in the operating theatre before the incision
  Arms: Placebo + Cefuroxime

SUMMARY:
During hysterectomy bacteria may enter into the peritoneal cavity through vaginal opening and contaminate the healing tissues. The risk for deep infection after hysterectomy is about 5%. By reducing post-hysterectomy infections, it is possible to reduce individual burden of disease in addition to the direct and indirect financial costs. This study primary aim is to assess if prophylactic preoperative use of azithromycin in addition to generally used cefuroxime decreases post-hysterectomy infections as compared to cefuroxime only prophylaxis during 30 days after hysterectomy. Secondary aim is to assess if there is change in post-hysterectomy superficial infections, urinary tract infections, or post-operative fever between the cohorts and to report possible side-effects of the used antibiotics. In addition, the study finds out a possible role of bacterial vaginosis and microbiome n post-hysterectomy infections.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing hysterectomy for benign indication in University Hospitals (Helsinki University Hospital, Turku University Hospital, Tampere University Hospital, Oulu University Hospital and Kuopio University Hospital) who have not any contraindications for azithromycin or cefuroxime.

Exclusion Criteria:

* Inability to understand the study protocol.
* Allergy for either cefuroxime or azithromycin.
* Congenital or acquired prolonged Q-T-corrected interval. All the participants will be asked about arrhythmias and whether they have congenital arrhythmias in the family,
* Electrocardiogram will be checked for all the participants.
* Use of medicines that may prolong Q-T-corrected interval (class Ia arrhythmia medications, quinidine, procainamide, and class III arrhythmia medications dofetilide, amiodarone and sotalol).
* Use of selective serotonin reuptake inhibitor medication and prolonged Q-T-corrected interval.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2278 (Estimated)
Dates: Start 2022-09-05 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Number of post-hysterectomy episodes with deep infections | Deep infections that occur between the first and 30th postoperative day after hysterectomy
  Number of deep wound and pelvic organ infection episodes reported by patients and doctors

SECONDARY OUTCOMES:
Number of other post-hysterectomy infections or fever episodes | Number of other infections or fever episodes that occur between the first and 30th postoperative day after hysterectomy.
  Number of superficial infections, other infections, such has urine tract infections, or fever episodes lasting over 38 ℃ over 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Päivi Rahkola-Soisalo, Adj prof, MD, Principal Investigator — Helsinki University Central Hospital; Tomi Mikkola, Prof, MD, Study Chair — Helsinki University Central Hospital; Päivi Rahkola-Soisalo, Adj prof, MD, Study Director — Helsinki University Central Hospital
Locations (6):
- Finland (6):
  - Helsinki University Central Hospital, Helsinki
  - Jyväskylä Central Hospital, Jyväskylä
  - Kuopio University Central Hospital, Kuopio
  - Oulu University Central Hospital, Oulu
  - Tampere University Central Hospital, Tampere
  - Turku University Central Hospital, Turku

IPD SHARING:
Plan to Share IPD: No